CLINICAL TRIAL: NCT01467050
Title: Prevention of Adverse Drug Events (ADEs) in Hospitalised Older Patients Using STOPP/START Criteria
Brief Title: Prevention of Adverse Drug Events (ADEs) in Hospitalised Older Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Denis O'Mahony, Senior Lecturer, Department of Medicine, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HRA_HSR/2010/14
Record Dates: First submitted 2011-08-31; First posted 2011-11-08 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Adverse Drug Reaction
Keywords: Adverse drug event; Adverse drug reaction; Inappropriate prescribing; Elderly; Hospital-acquired
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Potentially Inappropriate Medication List

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Application of STOPP/START criteria (Active Comparator)
  Interventions: Other: Application of STOPP/START criteria
- Control (No Intervention)
  Interventions: Other: Normal pharmaceutical care

INTERVENTIONS:
Other: Application of STOPP/START criteria — The researcher will apply the STOPP/START criteria to the cases randomised to this intervention. This will occur at the point of recruitment into the study and consists of applying STOPP/START criteria to the list of prescribed medications the patient is taking at that time point.
  Where potentially inappropriate medications (PIM's) are identified using the intervention, these are highlighted to the medical team with primary responsibility for the patient both verbally and in writing. The relevant registrar will be contacted in person or via telephone by the researcher and informed of the PIM's in addition to a standard medication advice form inserted into the patients' notes also highlighting the PIM's.
  Other Names: STOPP/START criteria for potentially inappropriate medications in older people.
  Arms: Application of STOPP/START criteria
Other: Normal pharmaceutical care — The normal process of medication prescription and review by the attending medical team.
  Arms: Control

SUMMARY:
The next four decades will see a marked expansion of the elderly population in Ireland, in particular people aged over 80 yrs. Persons aged over 80 are the highest consumers of prescription medicines in Ireland and have the highest prevalence rates of major polypharmacy. Polypharmacy is intimately linked with serious adverse drug events (ADEs) and consequent major morbidity and mortality. Epidemiological data from the United States indicate that ADEs is the fifth most common cause of death nationally. Experts suggest that effective evidence based interventions can be applied to this major public health problem.

Recent research data indicate a cause-and-effect relationship between inappropriate prescription medicines and serious ADEs in older people in hospital. To date, Beers' criteria have been the dominant set of criteria for defining potentially inappropriate medicines (PIMs) in late life. Research data collected by this group show that the recently validated STOPP/START criteria (Screening Tool of Older Persons' Prescriptions and Screening Tool to Alert doctors to Right Treatment) identify ADEs that are causal or contributory to acute hospital admission in older people 2.7 times more frequently than Beers' criteria. Based on these findings, our hypothesis is that STOPP/START criteria have the potential to be used as a regular intervention for the purpose of ADE prevention in older people. A recent single centre randomised control trial (RCT) undertaken at Cork University Hospital showed that prospective application of STOPP/START criteria led to a highly significant improvement in medication appropriateness in older hospitalised patients compared with standard inpatient pharmaceutical care. Significantly, the improvement in medication appropriateness was maintained to the end of the study follow-up i.e. 6 months post-discharge. However, the ability of STOPP/START criteria to significantly reduce ADEs in a prospective RCT has yet to be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 65 years and over presenting to CUH Accident and Emergency Departments with acute illness for admission under a medical or surgical team.

Exclusion Criteria:

1. Age less than 65 years.
2. Patient to be admitted under the care of a Geriatrician Psychiatrist of Old Age or Clinical Pharmacologist, or having been admitted under these services or attended their outpatient clinics in the previous 12 months. (These doctor groups are likely to minimise inappropriate medications in this population).
3. Terminally ill patient attended by palliative care team.
4. Critically ill patient e.g. admitted to Intensive Care Unit.
5. Patients who do not wish to participate in the study.
6. Patients whose hospital physician does not wish to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 732 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with probable and definite adverse drug events in hospital | Up to Day 14 of hospital admission

SECONDARY OUTCOMES:
drug ingredient cost at hospital discharge | Up to day 14
Composite health resource utilization including hospital readmissions and primary care consultations | At 3 months post discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Denis O'Mahony, MD, Principal Investigator — University College Cork, Ireland
Locations (1):
- Cork University Hospital, Cork, Munster, Ireland

REFERENCES:
- [Background] Gallagher PF, O'Connor MN, O'Mahony D. Prevention of potentially inappropriate prescribing for elderly patients: a randomized controlled trial using STOPP/START criteria. Clin Pharmacol Ther. 2011 Jun;89(6):845-54. doi: 10.1038/clpt.2011.44. Epub 2011 Apr 20. PMID 21508941
- [Background] O'Mahony D, Gallagher PF. Inappropriate prescribing in the older population: need for new criteria. Age Ageing. 2008 Mar;37(2):138-41. doi: 10.1093/ageing/afm189. PMID 18349010
- [Background] Hamilton H, Gallagher P, Ryan C, Byrne S, O'Mahony D. Potentially inappropriate medications defined by STOPP criteria and the risk of adverse drug events in older hospitalized patients. Arch Intern Med. 2011 Jun 13;171(11):1013-9. doi: 10.1001/archinternmed.2011.215. PMID 21670370
- [Background] Gallagher P, Ryan C, Byrne S, Kennedy J, O'Mahony D. STOPP (Screening Tool of Older Person's Prescriptions) and START (Screening Tool to Alert doctors to Right Treatment). Consensus validation. Int J Clin Pharmacol Ther. 2008 Feb;46(2):72-83. doi: 10.5414/cpp46072. PMID 18218287
- [Derived] O'Brien GL, O'Mahony D, Gillespie P, Mulcahy M, Walshe V, O'Connor MN, O'Sullivan D, Gallagher J, Byrne S. Cost-Effectiveness Analysis of a Physician-Implemented Medication Screening Tool in Older Hospitalised Patients in Ireland. Drugs Aging. 2018 Aug;35(8):751-762. doi: 10.1007/s40266-018-0564-0. PMID 30003429
- See also: Health Research Board of Ireland website — http://hrb.ie